CLINICAL TRIAL: NCT04595487
Title: Permanent Left Ventricular Septal Pacing Versus Right Ventricular Pacing in Patients With Atrioventricular Conduction Disorders: a Randomized Trial: LEAP Trial
Brief Title: LVSP vs RVP in Patients With AV Conduction Disorders
Acronym: LEAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL72047.068.20
Record Dates: First submitted 2020-10-01; First posted 2020-10-20 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Pacing; Pacing-Induced Cardiomyopathy; Conduction System Pacing; Left Ventricular Septal Pacing; Atrioventricular Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left ventricular septal pacing (Experimental): Implantation of a pacemaker with the ventricular lead delivered transvenously through the interventricular septum (IVS) to the left ventricular (LV) septum.
  Interventions: Procedure: Left ventricular septal pacing
- right ventricular pacing (Active Comparator): Implantation of a pacemaker with the ventricular lead placed in the RV.
  Interventions: Procedure: Right ventricular pacing

INTERVENTIONS:
Procedure: Left ventricular septal pacing — In the LVSP group, instead of placing the standard RV lead, the commercially available 3830 Select Secure (Medtronic, Minneapolis, USA) lead is introduced via standard transvenous approach and positioned against the right ventricular side of the IVS by using the commercially available non-deflectable septal delivery sheath (C315, Medtronic, Minneapolis, USA) under fluoroscopic guidance. Subsequently this pacing lead is advanced/screwed through the interventricular septum until the left ventricular septum is reached. Accurate lead position at the left ventricular septum will be determined anatomically using fluoroscopy, and electrically by evaluating local electrograms and changes in paced electrocardiogram morphology.
  In case of unsuccessful lead positioning in the left ventricular septum, the Select Secure lead may be placed at the His bundle region (natural conduction system of the heart) or in the right ventricle according to the physician's discretion.
  Arms: left ventricular septal pacing
Procedure: Right ventricular pacing — In the RVP group, the ventricular pacing lead is positioned in the right ventricle.
  Arms: right ventricular pacing

SUMMARY:
Rationale:

Permanent cardiac pacing is the only available therapy in patients with atrioventricular (AV) conduction disorders and can be life-saving. Right ventricular pacing (RVP), the routine clinical practice for decades in these patients, is non-physiologic, leads to dyssynchronous electrical and mechanical activation of the ventricles, and may cause pacing-induced cardiomyopathy and heart failure.

Left ventricular septal pacing (LVSP) is an emerging form of physiologic pacing that can possibly overcome the adverse effects of RVP.

Study design and hypotheses:

The LEAP trial is a multi-center investigator-initiated, prospective, randomized controlled, open label, blinded endpoint evaluation (PROBE) study that compares LVSP with conventional RVP. A total of four hundred seventy patients with a class I or IIa indication for pacemaker implantation due to AV conduction disorders and an expected ventricular pacing percentage >20% will be randomized 1:1 to LVSP or RVP. The primary endpoint is a composite endpoint of all-cause mortality, hospitalization for heart failure and a more than 10% decrease in left ventricular ejection fraction (LVEF) in absolute terms leading to a LVEF below 50% at one year follow-up. LVSP is anticipated to result in improved outcomes.

Secondary objectives are to evaluate whether LVSP is cost-effective and associated with an improved quality of life (QOL) as compared to RVP. Quality of life is expected to improve with LVSP and reduced healthcare resource utilizations are expected to ensure lower costs in the LVSP group during follow-up, despite initial higher costs of the implantation.

Study design: Multi-center investigator-initiated, prospective, randomized controlled, open label, blinded endpoint evaluation (PROBE) study.

Study population: Adult patients with a bradycardia-pacing indication because of AV conduction disorders with an expected ventricular pacing percentage of ≥ 20% and a left ventricular ejection fraction (LVEF) >/= 40%. Four hundred seventy patients will be randomized 1:1 to LVSP or RVP.

Intervention: LVSP vs RVP.

Main study parameters/endpoints:

The primary endpoint is a composite of all-cause mortality, hospitalization for heart failure, and a more than 10% point decrease in left ventricular ejection fraction (LVEF) leading to an LVEF below 50%, which as a binary combined endpoint will be determined at one year follow-up.

Secondary endpoints are:

* Time to first occurrence of all cause mortality or hospitalization for heart failure.
* Time to first occurrence of all cause mortality.
* Time to first occurrence of hospitalization for heart failure.
* Time to first occurrence of atrial fibrillation (AF) de novo.
* The echocardiographic changes in LVEF at one year.
* The echocardiographic changes in diastolic (dys-)function at one year.
* The occurrence of pacemaker related complications.
* Quality of life (QOL), cost-effectiveness analyses (CEA) and budget impact analysis (BIA).

The secondary endpoints (other than echocardiographic LVEF change) will be determined at the end of the follow-up period, when the last included patient has reached one year follow-up. The individual follow-up time for patients at this time point will vary with a minimum of one year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18y
* Life expectancy with good functional status of > 1y
* Class I or IIa pacemaker indication due to AV conduction disorder

  * Acquired 3rd or 2nd degree AVB
  * Atrial arrhythmia with slow ventricular conduction
* Expected ventricular pacing percentage > 20%
* LVEF >/= 40%
* Signed and dated informed consent form

Exclusion Criteria:

* HF NYHA class III-IV
* Class I indication for CRT
* Class I indication for ICD
* Previous implanted CIED (except for ILR)
* Atrial arrhythmia with planned AV junction ablation
* PCI or CABG <30 days before enrollment
* Valvular heart disease with indication for valve repair or replacement
* Hypertrophic cardiomyopathy with interventricular septum thickness > 2 cm
* Renal insufficiency requiring hemodialysis
* Active infectious disease or malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Binary combined endpoint consisting of all-cause mortality, hospitalization for heart failure, and a more than 10% point decrease in left ventricular ejection fraction (LVEF) leading to a LVEF below 50%. | Determined at one year follow-up
  Hospitalization for heart failure is defined as:
  1. hospitalization or unplanned hospital visits for heart failure requiring intravenous diuretics and/or (adjustment of) other medical heart failure therapy;
  2. hospitalization for upgrade to cardiac resynchronization therapy (CRT, ie biventricular pacing) for progression of heart failure with worsening NYHA class and/or (increased) need for diuretic therapy or other medical heart failure therapy;
  3. or hospitalization for upgrade to CRT for developing a class I indication for CRT (includes symptomatic heart failure);
  4. or hospitalization or unplanned hospital visit for heart failure triggered by an episode of atrial fibrillation with uncontrolled heart rate requiring intravenous diuretics or adjustment of rate control therapy.
  All-cause mortality is defined as death from any cause and subdivided into cardiovascular and non-cardiovascular death.

SECONDARY OUTCOMES:
Time to first occurrence of hospitalization for heart failure. | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  Hospitalization for heart failure is defined as:
  1. hospitalization or unplanned hospital visits for heart failure requiring intravenous diuretics and/or (adjustment of) other medical heart failure therapy;
  2. hospitalization for upgrade to cardiac resynchronization therapy (CRT, ie biventricular pacing) for progression of heart failure with worsening NYHA class and/or (increased) need for diuretic therapy or other medical heart failure therapy;
  3. or hospitalization for upgrade to CRT for developing a class I indication for CRT (includes symptomatic heart failure);
  4. or hospitalization or unplanned hospital visit for heart failure triggered by an episode of atrial fibrillation with uncontrolled heart rate requiring intravenous diuretics or adjustment of rate control therapy.
Time to first occurrence of all cause mortality. | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  All-cause mortality is defined as death from any cause and subdivided into cardiovascular and non-cardiovascular death.
Time to first occurrence of all cause mortality or hospitalization for heart failure. | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  All cause mortality and hospitalization for heart failure are defined as mentioned in secondary outcome 1 and 2.
Time to first occurrence of atrial fibrillation (AF) de novo. | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  Occurrence of atrial fibrillation de novo is defined as:
  Occurrence of a first clinical or subclinical episode of AF as diagnosed respectively by ECG (clinical AF) or by pacemaker interrogation (subclinical AF/atrial high rate episode, lasting > 24 hours) in patients without a history of AF.
The echocardiographic changes in left ventricular ejection fraction (LVEF) at one year. | Determined at one year follow-up
  Change in LVEF is based on echocardiography at one year follow-up as compared to baseline echocardiography.
The echocardiographic changes in diastolic (dys-)function at one year. | Determined at one year follow-up
  Diastolic function will be assessed by determining the following echocardiographic parameters at baseline and one year follow-up: E-wave, A-wave, E/A ratio, e' septal and lateral, E/e', 2D-strain of the left ventricle and atrium, pressure gradient across the tricuspid valve (dPTI) and volume of the left-atrium (LAVI). Diastolic function will be graded according to the current guidelines.
The occurrence of pacemaker related complications. | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  Pacemaker (implantation) related complications occurring during pacemaker implantation or during follow-up after pacemaker implantation consisting of: pneumothorax; cardiac tamponade; pocket hematoma requiring re-intervention; pacemaker infection; lead luxation, dislocation, or perforation requiring re-intervention; pacemaker and lead dysfunction during follow-up (elevated threshold/sensing issues/early battery depletion) requiring re-intervention.
Quality of Life analysis reported as Quality Adjusted Life Years (QALYs) | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  Quality of life will be analyzed using the EQ-5D-5L questionnaire at baseline, 6 and 12 months follow-up and every 6 months thereafter.
Cost effectiveness analysis (CEA) | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  A trial based economical evaluation from a societal perspective will be performed in accordance with the Dutch guidelines for economical evaluations in healthcare.
  Resource use will be measured from a societal perspective using data from case record forms and the Medical Consumption (MCQ) and Productivity loss (PCQ) questionnaires.
Budget Impact Analysis (BIA) | Determined at the end of the follow-up period (when the last-included patient reached the one year follow-up period)
  Budget impact analysis will be performed from a societal, health care provider and health care insurer perspective. The eligible population will be estimated based on national health care data.
  Costs of the intervention and heart failure costs will be included. Indirect costs will not be included. The time horizon will be 3 years. The expected uptake rate will be estimated based on a panel of experts (cardiologists, implementation specialist, patient representatives) and analyses will be performed for this expected uptake rate and several slightly higher and lower uptake rates. Uncertainties and scenarios will be discussed in a panel of experts as well and different scenarios will be analysed. Recommendations of the ISPOR task force are followed for all BIA calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Luermans, MD PhD, Principal Investigator — Department of Cardiology; Kevin Vernooy, MD PhD, Principal Investigator — Department of Cardiology
Locations (13):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - University Hospital Gent, Ghent
- University Hospital Kralovske Vinohrady, Prague, Czechia
- Policlinico Casilino, Rome, Italy
- Netherlands (6):
  - Maastricht University, Maastricht, Limburg
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Sint Antonius Ziekenhuis, Nieuwegein
- University Hospital Jaegellonian, Krakow, Poland
- Hospital Universitario y Politecnico La Fe, Valencia, Spain
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No